CLINICAL TRIAL: NCT05171816
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre Phase III Study of Olaparib Plus Abiraterone Relative to Placebo Plus Abiraterone as First-line Therapy in Men With Metastatic Castration-resistant Prostate Cancer (PROpel Study)
Brief Title: Study on Olaparib Plus Abiraterone as First-line Therapy in Men With Metastatic Castration-resistant Prostate Cancer (China Cohort)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D081SC00001Sub
Record Dates: First submitted 2021-12-20; First posted 2021-12-29 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer (mCRPC)
MeSH Terms: interventions — olaparib; Abiraterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- olaparib plus abiraterone (Experimental): Olaparib is available as a film-coated tablet containing 100 milligrams (mg) or 150 milligrams (mg) of olaparib. Subjects will be administered olaparib orally at a dose of 300 milligrams (mg) twice daily (bid). The initial dosage of 300 milligrams (mg) twice daily will be composed of 2 x 150 milligrams (mg) tablets per dose. The 100 milligrams (mg) and 150 milligrams (mg) tablets will be used to manage dose reductions during the study.
  Abiraterone acetate with prednisone or prednisolone will be sourced locally as commercially available materials. Subjects will be administered abiraterone orally at a dose of 1000 milligrams (mg) once daily, in combination with prednisone or prednisolone 5 milligrams (mg) administered orally twice daily.
  Interventions: Drug: olaparib; Drug: abiraterone acetate
- placebo plus abiraterone (Placebo Comparator): Placebo to match olaparib is available as a film-coated tablet in 100 milligrams (mg) or 150 milligrams (mg). Subjects will be administered placebo orally at a dose of 300 milligrams (mg) twice daily (bid). The initial dosage of 300 milligrams (mg) twice daily will be composed of 2 x 150 milligrams (mg) tablets per dose. The 100 milligrams (mg) and 150 milligrams (mg) tablets will be used to manage dose reductions during the study.
  Abiraterone acetate with prednisone or prednisolone will be sourced locally as commercially available materials. Subjects will be administered abiraterone orally at a dose of 1000 milligrams (mg) once daily, in combination with prednisone or prednisolone 5 milligrams (mg) administered orally twice daily.
  Interventions: Drug: abiraterone acetate

INTERVENTIONS:
Drug: olaparib — 300 mg (2 x 150 milligrams (mg) tablets) twice daily
  Other Names: Lynparza
  Arms: olaparib plus abiraterone
Drug: abiraterone acetate — 1000 milligrams (mg) once daily
  Other Names: Zytiga

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety (including evaluating side effects) of combination of olaparib and abiraterone versus placebo and abiraterone in patients with metastatic castration-resistant prostate cancer (mCRPC) who have received no prior cytotoxic chemotherapy or new hormonal agents (NHAs) at metastatic castration-resistant prostate cancer (mCRPC) stage.

DETAILED DESCRIPTION:
PROpel is a phase III study evaluating the efficacy, safety, and tolerability of olaparib versus placebo when given in addition to abiraterone to patients with metastatic castration-resistant prostate cancer (mCRPC) who have not received prior chemotherapy or new hormonal agents (NHAs) for metastatic castration-resistant prostate cancer (mCRPC) (first-line setting).

Approximately 720 patients globally were planned to be randomized in PROpel in a 1:1 ratio to treatment with either olaparib and abiraterone or placebo and abiraterone. Enrolment had completed with a total of 796 patients randomised. Following the completion of global enrolment, the China cohort will randomise approximately 108 additional patients at sites in China, also in a 1:1 ratio.

This cohort will enable standalone safety and efficacy analyses to support Chinese regulatory requirements. Patients from China will not be included in the Full Analysis Set for the global study analysis. In addition, all of the statistical analyses defined in this SAP will be performed using all patients randomised at sites in Asian countries (South Korea and Japan) excluding China, to be designated the Asian subgroup analysis.

Patients will receive oral treatment with olaparib 300 mg twice daily + abiraterone 1000 mg once daily or placebo twice daily + abiraterone 1000 mg once daily. Patients in both treatment groups will also receive either prednisone or prednisolone 5 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in the study protocol.
2. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
3. For inclusion in i) the optional exploratory genetic research and ii) the optional biomarker research, patients must fulfill the following criteria:

   * Provision of informed consent for genetic research prior to collection of sample.
   * Provision of informed consent for biomarker research prior to collection of sample.

   If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.
4. Patients must be ≥18 years of age (or ≥19 years of age in South Korea) at the time of signing the informed consent form. For patients enrolled in Japan who are <20 years of age, written informed consent should be obtained from the patient and from his legally acceptable representative.
5. Histologically or cytologically confirmed prostate adenocarcinoma.
6. Metastatic status defined as at least 1 documented metastatic lesion on either a bone scan or a computed tomography(CT)/ magnetic resonance imaging (MRI) scan.
7. First-line metastatic castration-resistant prostate cancer (mCRPC).
8. Ongoing androgen deprivation with gonadotropin-releasing hormone analogue or bilateral orchiectomy, with serum testosterone <50 nanograms per decilitre (ng/dL) (<2.0 nanomoles per litre (nmol/L)) within 28 days before randomisation. Patients receiving androgen deprivation therapy (ADT) at study entry should continue to do so throughout the study.
9. Candidate for abiraterone therapy with documented evidence of progressive disease.
10. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment.
11. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, with no deterioration over the previous 2 weeks.
12. The participant has, in the opinion of the investigator, a life expectancy of at least 6 months.
13. Prior to randomisation, sites must confirm availability of either an archival formalin fixed, paraffin embedded (FFPE) tumour tissue sample, or a new biopsy taken during the screening window, which meets the minimum pathology and sample requirements in order to enable homologous recombination repair (HRR) status subgroup analysis of the primary endpoint radiographic progression-free survival (rPFS). If there is not written confirmation of the availability of tumour tissue prior to randomisation, the patient is not eligible for the study.
14. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib+abiraterone when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

1. Has a known additional malignancy that has had progression or has required active treatment in the last 5 years.
2. Patients with myelodysplastic syndrome (MDS)/ acute myeloid leukaemia (AML) or with features suggestive of yelodysplastic syndrome (MDS)/ acute myeloid leukaemia (AML).
3. Clinically significant cardiovascular disease Association Class II-IV heart failure or cardiac ejection fraction measurement of <50% during screening as assessed by echocardiography or multigated acquisition scan.
4. Planned or scheduled cardiac surgery or percutaneous coronary intervention procedure.
5. Prior revascularisation procedure (significant coronary, carotid, or peripheral artery stenosis).
6. Uncontrolled hypertension (systolic blood pressure (BP) ≥160 millimeters of mercury (mmHg) or diastolic blood pressure (BP) ≥95 millimeters of mercury (mmHg)).
7. History of uncontrolled pituitary or adrenal dysfunction.
8. Active infection or other medical condition that would make prednisone/prednisolone use contraindicated.
9. Any chronic medical condition requiring a systemic dose of corticosteroid >10 milligrams (mg) prednisone/prednisolone per day.
10. Patients who are considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
11. Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAEs] grade >2) caused by previous cancer therapy, excluding alopecia.
12. Patients with brain metastases. A scan to confirm the absence of brain metastases is not required.
13. Patients with spinal cord compression are excluded unless they are considered to have received definitive treatment for this and have evidence of clinically stable disease for 4 weeks.
14. Patients who are unevaluable for both bone and soft tissue progression
15. Patients who are unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
16. Immunocompromised patients
17. Patients with known active hepatitis infection (ie, hepatitis B or C).
18. Any previous treatment with Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerase (PARP) inhibitor, including olaparib.
19. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment. Patients who receive palliative radiotherapy need to stop radiotherapy 1 week before randomisation.
20. Any previous exposure to a Cytochrome P450 (CYP) 17 (17α-hydroxylase/C17,20-lyase) inhibitor (eg, abiraterone, orteronel).
21. Concomitant use of known strong Cytochrome P450 (CYP) 3A inhibitors (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
22. Concomitant use of known strong Cytochrome P450 (CYP) 3A inducers (eg, phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine or St John's wort) or moderate Cytochrome P450 (CYP) 3A inducers (eg, bosentan, efavirenz or modafinil). The required period prior to starting study treatment is 5 weeks for phenobarbital and enzalutamide and 3 weeks for other agents.
23. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
24. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
25. Participation in another clinical study with an investigational product or investigational medical devices within 1 month of randomisation.
26. History of hypersensitivity to olaparib or abiraterone, any of the excipients of olaparib or abiraterone, or drugs with a similar chemical structure or class to olaparib or abiraterone.
27. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca and Merck staff and/or staff at the study site).
28. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
29. Previous randomisation in the present study.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2026-04-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Clarke, M.D., Principal Investigator — Christie Hospital Foundation Trust; Fred Saad, MD, Principal Investigator — University of Montreal Hospital Center
Locations (16):
- China (16):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Guizhou
  - Research Site, Henan
  - Research Site, Hubei
  - Research Site, Hunan
  - Research Site, Jilin
  - Research Site, Liaoning
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Sichuan
  - Research Site, Xi'an
  - Research Site, Zhejiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 108 patients were planned to be randomized in the study. Actually 162 patients were screened, and 110 patients were randomized successfully.
Groups:
- Olaparib 300 mg bd + Abiraterone 1000 mg qd: Patients receive oral treatment with olaparib 300mg twice daily in combination with abiraterone 1000mg once daily
- Placebo bd + Abiraterone 1000 mg qd: Patients receive oral treatment with placebo twice daily in combination with abiraterone 1000mg once daily.
Period: Overall Study
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Started | 54 | 56
Completed | 36 | 40
Not Completed | 18 | 16
Not completed — Death | 18 | 16

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.5 (8.2) | 68.9 (7.6) | 69.2 (7.9)
Age, Customized [Number; unit: Participants]
  <65 | 13 | 17 | 30
  >=65 | 41 | 39 | 80
Sex/Gender, Customized [Number; unit: Participants]
  Male | 54 | 56 | 110
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 0 | 0 | 0
  NOT HISPANIC OR LATINO | 54 | 56 | 110
  NOT REPORTED | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN | 54 | 56 | 110
Region of Enrollment [Number; unit: Participants]
  China | 54 | 56 | 110

OUTCOME MEASURES:

1. Primary Outcome: Radiological Progression Free Survival (rPFS)
Description: Radiological progression free survival is defined as the time from randomisation until the earlier date of radiological progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomised therapy or receives another anticancer therapy prior to progression.
  Per RECIST v1.1, progression is defined as the sum of TLs has a 20% and absolute ≥ 5mm increase from nadir, and/or unequivocal progression in any non target lesions, and/or any new lesion identified.
  Per PCWG3, progression on a bone scan is defined as 2 or more new lesions observed from the first visit after baseline compared to baseline, or from all other visits compared to first visit after baseline. A confirmatory scan is required.
Time Frame: Tumour imaging CT/MRI and bone scan were assessed every 8 weeks from randomisation to week 24 and then every 12 weeks until RECIST progression. Patients were followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Months | 14.75 [12.06 to 22.11] | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Other — Exploratory; p = 0.2592, Log Rank — Nominal p-value; The 2-sided p-value was calculated using the log-rank test stratified by metastases; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.83 to 2.48] — HR and CI calculated using Cox Proportional Hazards model, where a HR < 1 favours olaparib+abiraterone. Stratification factors are the same as those used in the stratified log-rank test

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from date of randomisation to death due to any cause regardless of whether the patient withdraws from randomised therapy or receives another anticancer therapy.
  The 22Jan2024 DCO is the final data cut-off for the OS analysis and therefore no further updates will be made.
Time Frame: Assessed every 12 weeks from randomisation until death or data cut-off. The endpoint was followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum.
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Months | 27.83 [27.83 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Other — Exploratory; p = 0.7251, Log Rank — Nominal p-value; The 2-sided p-value was calculated using the log-rank test stratified by metastases; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.57 to 2.29] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to First Subsequent Anticancer Therapy or Death (TFST)
Description: Time to first subsequent anticancer therapy (excluding radiotherapy) is defined as the time from randomisation to the earlier of start date of the first subsequent anti cancer therapy after discontinuation of randomised treatment or death from any cause.
Time Frame: Assessed from from randomization on 30 day follow-up after last dose of study medication and every 12 weeks after that until DCO. The endpoint was followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum.
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Months | 19.1 [15.4 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | 17.6 [10.6 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Other — Exploratory; p = 0.9715, Log Rank — Nominal p-value; The 2-sided p-value was calculated using the log-rank test stratified by metastases; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.60 to 1.64] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Pain Progression (TTPP)
Description: Time to pain progression is defined as time from randomisation to pain progression based on the Brief Pain Inventory-Short Form (BPI-SF) Item 3 "worst pain in 24 hours" (range 0-10, a higher score indicates worse pain) and opiate analgesic use (Analgesic quantification algorithm [AQA] score, range 0-7, a higher score indicates increased opioid use). For patients who are asymptomatic at baseline: A ≥2 point change from baseline in average (4-7 days) worst pain score observed at 2 consecutive visits or initiation of opioid use; For patients who are symptomatic at baseline: A ≥2 point change from baseline in average (4-7 days) worst pain score observed at 2 consecutive visits and an average worst pain score ≥4, and no decrease in average opioid use (≥1-point decrease in AQA score from a starting value of ≥2), or increase in opioid use (≥1-point increase, or ≥2-point increase if the starting value is 0) at 2 consecutive follow-up visits.
Time Frame: The BPI-SF and AQA were assessed on screening, day 1, day 15, day 29, day 43, day 57, day 71, and every 4 weeks after week 13 until DCO. The endpoint was followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum.
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Other — Exploratory; p = 0.4937, Log Rank — Nominal p-value; The 2-sided p-value was calculated using the log-rank test stratified by metastases; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.20 to 2.06] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Opiate Use
Description: Time to opiate use is defined as the time from date of randomisation to the date of first opiate use for cancer related pain.
Time Frame: Assessed on screening, days 1, 29, and 57, every 4 weeks after week 13, treatment discontinuation, and 30-day follow-up after last dose of study medication. Followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum.
Population: Randomised patients who are not on opiates at baseline
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 51 | 47
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Other — Exploratory; p = 0.4923, Log Rank — Nominal p-value; The 2-sided p-value was calculated using the log-rank test stratified by metastases; Hazard Ratio (HR) = 1.65, 95% CI 2-sided [0.61 to 4.87] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to a Symptomatic Skeletal-Related Event (SSRE)
Description: Time from date of randomisation to date of first symptomatic skeletal-related event as defined by any of the following or a combination:
  * Use of radiation therapy to prevent or relieve skeletal symptoms.
  * Occurrence of new symptomatic pathological bone fractures (vertebral or non-vertebral).
  * Occurrence of spinal cord compression.
  * Orthopaedic surgical intervention for bone metastasis.
Time Frame: Assessed at every visit from randomisation up to and including treatment discontinuation visit. The endpoint was followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum.
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events

7. Secondary Outcome: Time to Second Progression or Death (PFS2)
Description: The time to PFS2 is defined as the time from date of randomisation to date of second progression on next-line (immediately after study treatment) anticancer therapy or death, whichever occurs earlier.
Time Frame: Assessed from randomization every 12 weeks following the progression event used for PFS and the start of the next-line anticancer therapy. The endpoint was followed up for 479 days (approx 16 months) at minimum and 913 days (approx 30 months) at maximum.
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Months | 28.71 [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Other — Exploratory; p = 0.3407, Log Rank — Nominal p-value; The 2-sided p-value was calculated using the log-rank test stratified by metastases; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.63 to 3.39] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in BPI-SF Pain Severity and Pain Interference
Description: All BPI-SF pain items including "worst pain" are scored on a 0-10 numeric rating scale (NRS) with 0=No Pain and 10=Worst Pain Imaginable.
  The pain severity domain consists of 4 items (item #3, item #4, item #5, and item #6) which assess pain at its "worst," "least," "average," and "now" (current pain) respectively on the 11-point NRS. The overall pain severity score is calculated for each patient/visit as the mean of the individual non-missing items.
  The pain interference domain score is a mean of 7 items: general activity (item #9A), mood (item #9B), walking ability (item #9C), normal work (item #9D), relations with other people (item #9E), sleep (item #9F), and enjoyment of life (item #9G), each scored on an 11-point NRS from 0 (Does not interfere) to 10 (Completely interferes).
  BPI-SF worst pain, pain severity and pain interference score changes can be a minimum of -10 and a maximum of 10. A negative change from baseline value indicates improvement.
Time Frame: Assessed from date of first subject randomised: 23Jul2021 to data cut off (China DCO): 22Jan2024 (913 days). BPI-SF were completed by patients daily for 7 consecutive days every 4 weeks. Change from baseline is reported every 4 weeks until week 49.
Population: Full Analysis Set (FAS), only patients with baseline assessment and at least one post treatment assessment are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Score
  Change from baseline in BPI-SF worst pain - Week 5: number analyzed (Participants) | 41 | 47
  Change from baseline in BPI-SF worst pain - Week 5 | -0.70 [-1.25 to -0.15] | -0.66 [-1.13 to -0.19]
  Change from baseline in BPI-SF worst pain - Week 9: number analyzed (Participants) | 36 | 45
  Change from baseline in BPI-SF worst pain - Week 9 | -1.37 [-2.05 to -0.69] | -0.61 [-1.11 to -0.12]
  Change from baseline in BPI-SF worst pain - Week 13: number analyzed (Participants) | 35 | 44
  Change from baseline in BPI-SF worst pain - Week 13 | -1.42 [-2.16 to -0.69] | -0.35 [-0.69 to -0.01]
  Change from baseline in BPI-SF worst pain - Week 17: number analyzed (Participants) | 38 | 44
  Change from baseline in BPI-SF worst pain - Week 17 | -1.22 [-2.01 to -0.43] | -0.38 [-0.94 to 0.18]
  Change from baseline in BPI-SF worst pain - Week 21: number analyzed (Participants) | 36 | 38
  Change from baseline in BPI-SF worst pain - Week 21 | -1.06 [-1.71 to -0.40] | -0.63 [-1.20 to -0.06]
  Change from baseline in BPI-SF worst pain - Week 25: number analyzed (Participants) | 36 | 35
  Change from baseline in BPI-SF worst pain - Week 25 | -0.95 [-1.63 to -0.27] | -0.74 [-1.33 to -0.16]
  Change from baseline in BPI-SF worst pain - Week 29: number analyzed (Participants) | 33 | 33
  Change from baseline in BPI-SF worst pain - Week 29 | -1.24 [-1.88 to -0.60] | -0.26 [-0.84 to 0.33]
  Change from baseline in BPI-SF worst pain - Week 33: number analyzed (Participants) | 31 | 34
  Change from baseline in BPI-SF worst pain - Week 33 | -0.78 [-1.66 to 0.09] | -0.66 [-1.31 to -0.01]
  Change from baseline in BPI-SF worst pain - Week 37: number analyzed (Participants) | 30 | 32
  Change from baseline in BPI-SF worst pain - Week 37 | -0.61 [-1.25 to 0.03] | -0.59 [-1.19 to 0.02]
  Change from baseline in BPI-SF worst pain - Week 41: number analyzed (Participants) | 24 | 31
  Change from baseline in BPI-SF worst pain - Week 41 | -0.10 [-1.09 to 0.88] | -0.43 [-0.97 to 0.10]
  Change from baseline in BPI-SF worst pain - Week 45: number analyzed (Participants) | 26 | 30
  Change from baseline in BPI-SF worst pain - Week 45 | -0.46 [-1.47 to 0.56] | -0.19 [-0.74 to 0.36]
  Change from baseline in BPI-SF worst pain - Week 49: number analyzed (Participants) | 24 | 27
  Change from baseline in BPI-SF worst pain - Week 49 | 0.11 [-0.81 to 1.02] | -0.06 [-0.59 to 0.47]
  Change from baseline in BPI-SF overall pain severity score - Week 5: number analyzed (Participants) | 41 | 47
  Change from baseline in BPI-SF overall pain severity score - Week 5 | -0.51 [-0.98 to -0.05] | -0.56 [-0.98 to -0.13]
  Change from baseline in BPI-SF overall pain severity score - Week 9: number analyzed (Participants) | 36 | 45
  Change from baseline in BPI-SF overall pain severity score - Week 9 | -1.12 [-1.65 to -0.60] | -0.54 [-1.00 to -0.08]
  Change from baseline in BPI-SF overall pain severity score - Week 13: number analyzed (Participants) | 35 | 44
  Change from baseline in BPI-SF overall pain severity score - Week 13 | -1.21 [-1.78 to -0.63] | -0.31 [-0.60 to -0.02]
  Change from baseline in BPI-SF overall pain severity score - Week 17: number analyzed (Participants) | 38 | 44
  Change from baseline in BPI-SF overall pain severity score - Week 17 | -1.02 [-1.67 to -0.38] | -0.34 [-0.85 to 0.16]
  Change from baseline in BPI-SF overall pain severity score - Week 21: number analyzed (Participants) | 36 | 38
  Change from baseline in BPI-SF overall pain severity score - Week 21 | -0.87 [-1.39 to -0.35] | -0.57 [-1.09 to -0.06]
  Change from baseline in BPI-SF overall pain severity score - Week 25: number analyzed (Participants) | 36 | 35
  Change from baseline in BPI-SF overall pain severity score - Week 25 | -0.81 [-1.37 to -0.25] | -0.68 [-1.22 to -0.14]
  Change from baseline in BPI-SF overall pain severity score - Week 29: number analyzed (Participants) | 33 | 33
  Change from baseline in BPI-SF overall pain severity score - Week 29 | -0.94 [-1.46 to -0.42] | -0.26 [-0.71 to 0.18]
  Change from baseline in BPI-SF overall pain severity score - Week 33: number analyzed (Participants) | 31 | 34
  Change from baseline in BPI-SF overall pain severity score - Week 33 | -0.72 [-1.36 to -0.08] | -0.63 [-1.20 to -0.06]
  Change from baseline in BPI-SF overall pain severity score - Week 37: number analyzed (Participants) | 30 | 32
  Change from baseline in BPI-SF overall pain severity score - Week 37 | -0.43 [-0.90 to 0.03] | -0.51 [-0.94 to -0.08]
  Change from baseline in BPI-SF overall pain severity score - Week 41: number analyzed (Participants) | 24 | 31
  Change from baseline in BPI-SF overall pain severity score - Week 41 | -0.19 [-0.74 to 0.36] | -0.42 [-0.83 to -0.01]
  Change from baseline in BPI-SF overall pain severity score - Week 45: number analyzed (Participants) | 26 | 30
  Change from baseline in BPI-SF overall pain severity score - Week 45 | -0.45 [-1.12 to 0.22] | -0.26 [-0.65 to 0.12]
  Change from baseline in BPI-SF overall pain severity score - Week 49: number analyzed (Participants) | 24 | 27
  Change from baseline in BPI-SF overall pain severity score - Week 49 | -0.01 [-0.52 to 0.50] | -0.21 [-0.64 to 0.21]
  Change from baseline in BPI-SF overall pain interference score - Week 5: number analyzed (Participants) | 41 | 47
  Change from baseline in BPI-SF overall pain interference score - Week 5 | -0.21 [-0.75 to 0.33] | -0.30 [-0.71 to 0.12]
  Change from baseline in BPI-SF overall pain interference score - Week 9: number analyzed (Participants) | 36 | 45
  Change from baseline in BPI-SF overall pain interference score - Week 9 | -0.88 [-1.41 to -0.35] | -0.33 [-0.83 to 0.17]
  Change from baseline in BPI-SF overall pain interference score - Week 13: number analyzed (Participants) | 35 | 44
  Change from baseline in BPI-SF overall pain interference score - Week 13 | -0.98 [-1.53 to -0.42] | -0.14 [-0.44 to 0.15]
  Change from baseline in BPI-SF overall pain interference score - Week 17: number analyzed (Participants) | 38 | 44
  Change from baseline in BPI-SF overall pain interference score - Week 17 | -0.83 [-1.47 to -0.19] | -0.16 [-0.68 to 0.37]
  Change from baseline in BPI-SF overall pain interference score - Week 21: number analyzed (Participants) | 36 | 38
  Change from baseline in BPI-SF overall pain interference score - Week 21 | -0.70 [-1.24 to -0.15] | -0.31 [-0.84 to 0.21]
  Change from baseline in BPI-SF overall pain interference score - Week 25: number analyzed (Participants) | 36 | 35
  Change from baseline in BPI-SF overall pain interference score - Week 25 | -0.53 [-1.14 to 0.09] | -0.42 [-0.97 to 0.13]
  Change from baseline in BPI-SF overall pain interference score - Week 29: number analyzed (Participants) | 33 | 33
  Change from baseline in BPI-SF overall pain interference score - Week 29 | -0.78 [-1.33 to -0.23] | 0.02 [-0.37 to 0.42]
  Change from baseline in BPI-SF overall pain interference score - Week 33: number analyzed (Participants) | 31 | 34
  Change from baseline in BPI-SF overall pain interference score - Week 33 | -0.70 [-1.43 to 0.03] | -0.35 [-0.94 to 0.24]
  Change from baseline in BPI-SF overall pain interference score - Week 37: number analyzed (Participants) | 30 | 32
  Change from baseline in BPI-SF overall pain interference score - Week 37 | -0.21 [-0.68 to 0.26] | -0.09 [-0.50 to 0.31]
  Change from baseline in BPI-SF overall pain interference score - Week 41: number analyzed (Participants) | 24 | 31
  Change from baseline in BPI-SF overall pain interference score - Week 41 | -0.05 [-0.59 to 0.49] | -0.18 [-0.57 to 0.21]
  Change from baseline in BPI-SF overall pain interference score - Week 45: number analyzed (Participants) | 26 | 30
  Change from baseline in BPI-SF overall pain interference score - Week 45 | -0.36 [-1.01 to 0.30] | -0.13 [-0.52 to 0.26]
  Change from baseline in BPI-SF overall pain interference score - Week 49: number analyzed (Participants) | 24 | 27
  Change from baseline in BPI-SF overall pain interference score - Week 49 | 0.09 [-0.39 to 0.57] | -0.15 [-0.56 to 0.26]

9. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy- Prostate Cancer (FACT-P)
Description: The following measures are calculated from the FACT-P questionnaire, the resulting value is the total score for the associated questions or scaled scores:
  * Physical well-being subscale (PWB) (Questions GP1 to GP7)
  * Social/family well-being subscale (SWB) (Questions GS1 to GS7)
  * Emotional well-being subscale (EWB) (Questions GE1 to GE6)
  * Functional well-being subscale (FWB) (Questions GF1 to GF7)
  * Prostate cancer subscale (PCS) (Questions C2, C6, P1 to P8, BL2 and BL5) The scores range from 0 ("Not at all") to 4 ("Very much") for positively phrased questions, and from 0 ("Very much") to 4 ("Not at all") for negatively phrased questions.
  Total FACT-P score is the sum of PWB, SWB, EWB, FWB and PCS. FACT-P total score changes can be a minimum of -156 and a maximum of 156. A positive value indicates improvement.
  FACT-G total score is the sum of PWB, SWB, EWB and FWB. FACT-G Total score changes can be a minimum of -108 and a maximum of 108. A positive value indicates improvement.
Time Frame: Assessed from date of first subject randomised: 23Jul2021 to data cut off (China DCO): 22Jan2024 (913 days). FACT-P were assessed every 4 weeks from Day 1 until Week 52. Change from baseline is reported every 4 weeks until week 49.
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 54 | 56
Score
  Change from baseline in FACT-P Total - Week 5: number analyzed (Participants) | 38 | 46
  Change from baseline in FACT-P Total - Week 5 | -4.43 [-11.40 to 2.54] | -0.84 [-4.92 to 3.25]
  Change from baseline in FACT-P Total - Week 9: number analyzed (Participants) | 35 | 43
  Change from baseline in FACT-P Total - Week 9 | -4.95 [-12.69 to 2.79] | 1.00 [-4.80 to 6.79]
  Change from baseline in FACT-P Total - Week 13: number analyzed (Participants) | 36 | 43
  Change from baseline in FACT-P Total - Week 13 | -1.51 [-7.95 to 4.92] | -3.07 [-8.49 to 2.36]
  Change from baseline in FACT-P Total - Week 17: number analyzed (Participants) | 35 | 42
  Change from baseline in FACT-P Total - Week 17 | -1.82 [-10.00 to 6.36] | -3.51 [-9.63 to 2.60]
  Change from baseline in FACT-P Total - Week 21: number analyzed (Participants) | 35 | 37
  Change from baseline in FACT-P Total - Week 21 | -6.60 [-15.08 to 1.88] | -0.54 [-7.07 to 6.00]
  Change from baseline in FACT-P Total - Week 25: number analyzed (Participants) | 34 | 35
  Change from baseline in FACT-P Total - Week 25 | -6.55 [-16.46 to 3.36] | -1.68 [-8.30 to 4.95]
  Change from baseline in FACT-P Total - Week 29: number analyzed (Participants) | 31 | 35
  Change from baseline in FACT-P Total - Week 29 | -1.32 [-11.86 to 9.22] | 0.62 [-6.28 to 7.53]
  Change from baseline in FACT-P Total - Week 33: number analyzed (Participants) | 28 | 34
  Change from baseline in FACT-P Total - Week 33 | -7.23 [-17.13 to 2.68] | -0.75 [-6.97 to 5.46]
  Change from baseline in FACT-P Total - Week 37: number analyzed (Participants) | 26 | 33
  Change from baseline in FACT-P Total - Week 37 | -3.21 [-11.48 to 5.07] | -4.87 [-11.95 to 2.22]
  Change from baseline in FACT-P Total - Week 41: number analyzed (Participants) | 25 | 31
  Change from baseline in FACT-P Total - Week 41 | -7.16 [-15.95 to 1.63] | 0.47 [-6.04 to 6.99]
  Change from baseline in FACT-P Total - Week 45: number analyzed (Participants) | 24 | 31
  Change from baseline in FACT-P Total - Week 45 | -8.28 [-17.49 to 0.92] | -1.69 [-7.76 to 4.39]
  Change from baseline in FACT-P Total - Week 49: number analyzed (Participants) | 23 | 26
  Change from baseline in FACT-P Total - Week 49 | -9.78 [-17.36 to -2.21] | -1.35 [-6.72 to 4.02]
  Change from baseline in FACT-G Total - Week 5: number analyzed (Participants) | 38 | 46
  Change from baseline in FACT-G Total - Week 5 | -4.85 [-9.84 to 0.14] | -1.75 [-4.92 to 1.42]
  Change from baseline in FACT-G Total - Week 9: number analyzed (Participants) | 35 | 43
  Change from baseline in FACT-G Total - Week 9 | -4.55 [-10.27 to 1.17] | -0.07 [-3.80 to 3.66]
  Change from baseline in FACT-G Total - Week 13: number analyzed (Participants) | 36 | 43
  Change from baseline in FACT-G Total - Week 13 | -2.43 [-6.97 to 2.11] | -3.79 [-7.41 to -0.16]
  Change from baseline in FACT-G Total - Week 17: number analyzed (Participants) | 35 | 42
  Change from baseline in FACT-G Total - Week 17 | -2.45 [-8.19 to 3.29] | -4.30 [-7.98 to -0.62]
  Change from baseline in FACT-G Total - Week 21: number analyzed (Participants) | 35 | 37
  Change from baseline in FACT-G Total - Week 21 | -5.26 [-11.49 to 0.98] | -2.10 [-6.40 to 2.20]
  Change from baseline in FACT-G Total - Week 25: number analyzed (Participants) | 34 | 35
  Change from baseline in FACT-G Total - Week 25 | -6.23 [-13.50 to 1.04] | -3.45 [-8.39 to 1.49]
  Change from baseline in FACT-G Total - Week 29: number analyzed (Participants) | 31 | 35
  Change from baseline in FACT-G Total - Week 29 | -2.26 [-10.15 to 5.63] | -1.35 [-6.27 to 3.57]
  Change from baseline in FACT-G Total - Week 33: number analyzed (Participants) | 28 | 34
  Change from baseline in FACT-G Total - Week 33 | -6.15 [-13.40 to 1.09] | -2.75 [-7.38 to 1.87]
  Change from baseline in FACT-G Total - Week 37: number analyzed (Participants) | 26 | 33
  Change from baseline in FACT-G Total - Week 37 | -1.32 [-7.26 to 4.62] | -5.14 [-10.32 to 0.04]
  Change from baseline in FACT-G Total - Week 41: number analyzed (Participants) | 25 | 31
  Change from baseline in FACT-G Total - Week 41 | -5.72 [-12.30 to 0.86] | -1.08 [-5.90 to 3.75]
  Change from baseline in FACT-G Total - Week 45: number analyzed (Participants) | 24 | 31
  Change from baseline in FACT-G Total - Week 45 | -5.70 [-12.48 to 1.08] | -2.27 [-6.78 to 2.24]
  Change from baseline in FACT-G Total - Week 49: number analyzed (Participants) | 23 | 26
  Change from baseline in FACT-G Total - Week 49 | -7.78 [-13.34 to -2.22] | -1.51 [-5.13 to 2.11]

ADVERSE EVENTS:
Time Frame: Adverse events with an onset date, or worsen, on or after the date of first dose and up to and including 30 days following discontinuation of randomised treatment. Assessed from date of randomisation to data cut off (China DCO): 22Jan2024 (Approx. 2 years 7 months)
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
All-Cause Mortality (participants affected / at risk) | 18/54 | 16/56
Serious Adverse Events (participants affected / at risk) | 23/54 | 21/56
Other Adverse Events (participants affected / at risk) | 53/54 | 54/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd + Abiraterone 1000 mg qd (N=54) | Placebo bd + Abiraterone 1000 mg qd (N=56)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd + Abiraterone 1000 mg qd (N=54) | Placebo bd + Abiraterone 1000 mg qd (N=56)
Chronic gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (12) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 42 (78) | 18 (29)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (4)
Asthenia (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 4 (5) | 4 (4)
Oedema peripheral (General disorders) | 4 (5) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 3 (8)
Covid-19 (Infections and infestations) | 5 (5) | 7 (7)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Suspected covid-19 (Infections and infestations) | 3 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Alanine aminotransferase increased (Investigations) | 11 (18) | 14 (21)
Amylase increased (Investigations) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 11 (18) | 11 (16)
Bile acids increased (Investigations) | 1 (3) | 7 (10)
Blood alkaline phosphatase increased (Investigations) | 9 (13) | 5 (5)
Blood bilirubin increased (Investigations) | 14 (29) | 15 (27)
Blood bilirubin unconjugated increased (Investigations) | 3 (4) | 0 (0)
Blood creatinine increased (Investigations) | 7 (18) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 4 (4)
Electrocardiogram st segment abnormal (Investigations) | 1 (1) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 5 (6) | 2 (2)
Lymphocyte count decreased (Investigations) | 13 (24) | 5 (10)
Neutrophil count decreased (Investigations) | 10 (14) | 1 (2)
Neutrophil count increased (Investigations) | 1 (1) | 3 (5)
Platelet count decreased (Investigations) | 8 (19) | 5 (7)
Weight decreased (Investigations) | 10 (15) | 6 (8)
Weight increased (Investigations) | 4 (4) | 3 (3)
White blood cell count decreased (Investigations) | 11 (25) | 3 (8)
White blood cell count increased (Investigations) | 1 (1) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 6 (12) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 (20) | 12 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (17) | 11 (18)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (18) | 13 (20)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 (28) | 11 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (9) | 5 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 3 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (14) | 13 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 6 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 3 (4)
Renal impairment (Renal and urinary disorders) | 8 (17) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 5 (6)
Hypertension (Vascular disorders) | 3 (5) | 7 (9)

LIMITATIONS AND CAVEATS:
The study treatment period overlapped with the COVID-19 global pandemic caused by SARS-CoV-2 and declared by the World Health Organization on 11 March 2020. 55 patients had a visit impacted by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT05171816/Prot_008.pdf
  • Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT05171816/SAP_009.pdf